CLINICAL TRIAL: NCT01794416
Title: Thoracoscopic Ablation Versus Endocardial Ablation in Patient With Paroxysmal Atrial Fibrillation After Failed Initial Endocardial Ablation
Brief Title: Thoracoscopic Versus Endocardial Ablation in Patient With Paroxysmal AF After Failed Initial Endocardial Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-EA-001
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracoscopic epicardial ablation (Active Comparator): Patients were treated with video-assisted thoracoscopy under general anesthesia. PVI was performed from the epicardial side with a bipolar RF ablation clamp (AtriCure). At least 2 overlapping applications around each of the ipsilateral veins were made, and isolation was confirmed by the absence of PV potentials and exit block during pacing. An additional application was made in the interatrial Waterston groove in the right side to isolate the ganglionic plexi from the atria. On the left side, the ligament of Marshal was cut, but no additional ablation of ganglionic plexi was pursued.
  The RevealXT (implantable loop recorder) was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.
  Interventions: Procedure: Thoracoscopic epicardial ablation; Device: Implantable loop recorder
- Endocardial catheter ablation (Active Comparator): Externally-irrigated tip (5-mm tip, Celsius Thermo-Cool, Biosense Webster, Diamond Bar, CA, USA). Temperature-controlled RF delivery was performed with a maximum power output of 50 W and temperature limit of 50 C. The catheter was irrigated using 0.9% saline infusion at a ﬂow rate of 20-40 mL/min during RF delivery and 2 mL/min between applications using a commercially available pump (Cool Flow, Biosense Webster). The RevealXT (implantable loop recorder) was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.
  Interventions: Procedure: Endocardial catheter ablation; Device: Implantable loop recorder

INTERVENTIONS:
Procedure: Thoracoscopic epicardial ablation
  Arms: Thoracoscopic epicardial ablation
Procedure: Endocardial catheter ablation
  Arms: Endocardial catheter ablation
Device: Implantable loop recorder

SUMMARY:
The investigators aimed to compare two approaches thoracoscopic epicardial ablation and endocardial catheter ablation after failed initial catheter ablation in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* failed initial catheter ablation
* paroxysmal atrial fibrillation

Exclusion Criteria:

* chronic lung disease
* body mass index >35
* longstanding atrial fibrillation 1 year
* previous stroke or transient ischemic attack
* left atrial thrombus
* left atrial size >65 mm
* left ventricular ejection fraction <35%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
freedom from any atrial arrhythmia | 12 months

SECONDARY OUTCOMES:
rate of significant adverse events (SAEs) | 12 months
atrial fibrillation burden by ILR | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Pokushalov E, Romanov A, Elesin D, Bogachev-Prokophiev A, Losik D, Bairamova S, Karaskov A, Steinberg JS. Catheter versus surgical ablation of atrial fibrillation after a failed initial pulmonary vein isolation procedure: a randomized controlled trial. J Cardiovasc Electrophysiol. 2013 Dec;24(12):1338-43. doi: 10.1111/jce.12245. Epub 2013 Sep 9. PMID 24016147
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru